CLINICAL TRIAL: NCT05864404
Title: Comparison of Patients' Satisfaction Between Dexmedetomidine and Remimazolam Anesthesia in Patients With Atrial Fibrillation Undergoing Catheter Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 4-2023-0173
Record Dates: First submitted 2023-04-18; First posted 2023-05-18 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Patients With Atrial Fibrillation Undergoing Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam-remifentanil (RR group) (Experimental)
  Interventions: Drug: remimazolam-remifentanil
- dexmedetomidine-remifentanil (DR group) (Active Comparator)
  Interventions: Drug: dexmedetomidine-remifentanil

INTERVENTIONS:
Drug: remimazolam-remifentanil — In the case of remimazolam, the bolus is prepared in a 30cc syringe by mixing 0.075mg/kg and normal saline to make a total of 25mL. Inject the bolus at a rate of 150 cc/h, and measure the sedation depth every 2 to 3 minutes, stopping the infusion when the target sedation depth (RASS -1 to -2 points) is reached. Remimazolam is then infused at 0.5 to 1 mg/kg/hr to maintain the target depth of sedation until the end of the procedure. Remifentanil was infused at a rate of 1.2-7.2 mcg/kg/h.
  Arms: remimazolam-remifentanil (RR group)
Drug: dexmedetomidine-remifentanil — In the case of dexmedetomidine, the bolus is prepared in a 30cc syringe by mixing 1.0mcg/kg and normal saline to make a total of 25mL. Inject the bolus at a rate of 150 cc/h, and measure the sedation depth every 2 to 3 minutes, stopping the infusion when the target sedation depth (RASS -1 to -2 points) is reached. Dexmedetomidine is then infused at 0.4 to 0.8 mcg/kg/h to maintain the target depth of sedation until the end of the procedure. Remifentanil was infused at a rate of 1.2-7.2 mcg/kg/h.
  Arms: dexmedetomidine-remifentanil (DR group)

SUMMARY:
The primary purpose of this study was to investigate whether remimazolam administration for sedation had a positive effect on patients' satisfaction compared to dexmedetomidine administration in patients with atrial fibrillation undergoing catheter ablation.

Atrial fibrillation is a common arrhythmia in clinical practice. Catheter ablation can be used when the cause of atrial fibrillation is in the pulmonary veins. However, the procedure takes 2 to 4 hours, and patients complain of considerable discomfort. Remimazolam has the advantage of having no drug interaction with CYP3A4 and shorter elimination half-life, duration of action, and shorter recovery time than midazolam, a previously used drug. In addition, compared to dexmedetomidine, side effects such as bradycardia and hypotension are expected to be less. In addition, even if unexpected deep sedation is induced, complete reversal using flumazenil is possible, so the risk of re-sedation could be low.

In other words, when remimazolam is used instead of a drug previously used as a sedative in atrial fibrillation patients undergoing catheter ablation, effects such as rapid action and recovery, reduced complications, improved safety, and improved patient satisfaction can be expected. Therefore, this study was designed to confirm the hypothesis that administration of remimazolam would improve satisfaction in patients undergoing catheter ablation compared to dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-79 years, gender not limited
* Patients undergoing catheter ablation for atrial fibrillation who require monitored anesthetic care (MAC).
* Patients with an American Society of Anesthesiologists (ASA) physical status classification 1,2,3.

Exclusion Criteria:

* Patients with an American Society of Anesthesiologists (ASA) physical status classification >3.
* Patients with a history of psychiatric disorders
* Patients with myocardial infarction or stroke within the past year
* Patients with a history of major vascular surgery or cardiac surgery within the past year
* Patients with reduced liver function, chronic kidney disease (stage 3 or higher)
* Patients diagnosed with heart failure with a left ventricular ejection fraction <40%
* Patients who need vasopressor or oxygen therapy due to unstable vital signs before procedure.
* Patients with fever (>38°) or severe uncontrolled high blood pressure
* Patients with a history of drug hypersensitivity during previous anesthesia
* Patients who are unable to communicate and have cognitive impairment
* Patients with a history of drug or alcohol addiction
* Patients with a history of obstructive sleep apnea

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-10-09 (Estimated); Study Completion 2024-10-09 (Estimated)

PRIMARY OUTCOMES:
The satisfaction levels of the patients | Immediately after the procedure
  The satisfaction levels of the patients was assessed with a 5-point numerical scale (0=extremely dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, and 4=extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided